Study Title: Prospective, open-label trial to evaluate efficacy of 30-day

duration of fidaxomicin in patients with recurrent Clostridioides

(Clostridium) difficile infection.

**Protocol Version Date/Number** 01OCT2020 Version No. 5

ClinicalTrial.gov NCT02395848

Protocol No: CDI.FIDAXOMICIN.1

**Primary Investigator Name:** Christine H. Lee

Primary Investigator Address: Vancouver Island Health Authority 1952 Bay Street. Victoria, BC

V8R 1J8

Safety Reporting: Vancouver Island Health Authority Clinical Research Ethics Board

## 1 STUDY RATIONALE/BACKGROUND

Clostridioides difficile (C. difficile) infection (CDI) is one of the most frequent causes of healthcare associated infections and its rates are also growing in the community. The case fatality rate associated with CDI is 6%. CDI is also problematic as it can lead to chronic diarrhea and has been the source of outbreaks in many hospitals. 1-6

The efficacy of standard antibiotics especially for recurrent CDI is limited as oral vancomycin and metronidazole also suppress the growth of anaerobic bacteria such as *Bacteroides fragilis* (*B. fragilis*) group which protect against proliferation of *C. difficile*. In contrast, in vitro study has shown that fidaxomicin has negligible activity against *B. fragilis*. The persistent disruption of healthy colonic flora may be the reason for recurrences following a course of treatment with metronidazole or vancomycin. Fidaxomicin has shown to reduce recurrences by approximately 50% when compared to oral vancomycin for primary or 1<sup>st</sup> episode of recurrent CDI.

There is a growing concern regarding failure rates for metronidazole, which is recommended as the first line therapy for uncomplicated CDI; as it has risen from 2.5% to greater than 18% since 2000.¹ Recurrence of CDI following a course of standard antibiotic (metronidazole/oral vancomycin) therapy is high, especially in the elderly patients over 65 years of age, in hospitalized and in the immunocompromised patients. Rates of recurrences are greater than 50% for those over the age 65.9 The risk of further recurrence is over 60% for patients who have failed 3 or more episodes of standard antimicrobial therapies.9-12 Fecal microbiota transplantation (FMT) has shown to be very effective for multiple recurrent CDI.¹ Although effective, FMT has limitations as the majority of healthcare facilities, worldwide do not have the infrastructure available to offer the treatment as it requires readily available donors and laboratory capacity to screen donors and manufacture FMT in timely manner. There are also potential risks associated with FMT such as transmission of pathogens, including SARS-CoV-2, antibiotic resistant organism, development of bacteremia especially in immunocompromised hosts, peritonitis and intestinal perforation. 14-16

Determining the efficacy and safety of 30-day duration of fidaxomicin for recurrent CDI through an open label clinical trial has important implications for policy making related to the drug reimbursement programs. In addition, the results of this study will be instrumental in demonstrating to the scientific and healthcare communities there may be a role for the 30-day

Protocol No: CDI.FIDAXOMICIN.1 Version No. 5
Date: 01OCT2020 

course of fidaxomicin as a treatment modality for recurrent CDI. Curing CDI will restore the health and quality of life not just at the individual patient level but to the healthcare communities as well. Patients with refractory CDI require prolonged hospital admission, which increases the organism burden within the healthcare facilities. This in turn leads to the spread of the infection to other vulnerable patients. If a 30-day course of fidaxomicin proves to be safe and effective in curing patients with recurrent CDI, it will reduce the risk of severe complications in each patient and reduce transmission of CDI to other susceptible patients. All these will also reduce healthcare costs.

# 2 STUDY HYPOTHESIS

Thirty-day duration of fidaxomicin will be effective in reducing the rates of recurrence of CDI. Fidaxomicin has shown to reduce recurrences by 50% when compared to oral vancomycin for primary or 1<sup>st</sup> episode of recurrent CDI. In vitro study has shown that fidaxomicin has virtually no activity against *B. fragilis* and may explain the significant reduction in *C. difficile* recurrences.

# 3 STUDY OBJECTIVE AND ENDPOINTS

# 3.1 STUDY OBJECTIVE

To study the outcome of patients treated with a 30-day course of fidaxomicin for recurrent CDI

#### 3.2 STUDY ENDPOINTS

## 3.2.1 PRIMARY EFFICACY ENDPOINT

- 1. Clinical response at study day 30, in this context, clinical response will be defined as those participants who have improvement in the number of bowel movements as determined by  $\leq 3$  unformed stools in a 24-hour period for 2 consecutive days during treatment and remaining well through study day 30.
- 2. Sustained clinical response as defined by those participants who achieved clinical response by study day 30 and did not experience a recurrence of CDI at the end of the follow-up period, evaluated at 8 weeks after the completion of treatment.
- 3. Recurrence of CDI as defined by return of diarrhea (a minimum of 3 unformed bowel movements or ≥ 200 mL of stool for individuals with a stool collection device such as rectal tube or colostomy within a 24-hour period) and positive stool test after a period of symptom resolution within study period and has received at least a 10-day course of standard antibiotic therapy.
- 4. Treatment failure as defined by patients not meeting the definition of cure and requiring additional treatment(s) for current CDI episode.

## 3.2.2 **SECONDARY ENDPOINT(S)**:

- The evaluation of safety of 30-day duration of fidaxomicin (200mg twice daily x 10 days and 200mg once daily x 20 days).
  - O Assessment for adverse reactions by history, complete blood count and chemistry panel at day 10 (-3, +1d), followed by history on day 30 (+/-3d) and week 8 post treatment (week 12) of the study period.
- Any serious adverse events up to and including week 12 for any of the following:
  - o Death or a life-threatening event
  - New hospitalization or prolongation of current hospitalization
  - o A significant new incapacity to conduct normal life functions

Date: 01OCT2020 

# 4 STUDY DESIGN

#### 4.1 SITES

Vancouver Island Health Authority

## 4.2 INCLUSION/EXCLUSION CRITERIA

## 4.2.1 INCLUSION CRITERIA

- 1. Age 18 years or older.
- 2. Able to provide informed consent.
- 3. Willing and able to comply with all the required study procedures.
- 4. A positive stool test for *C. difficile* toxin/gene using either PCR or enzyme immunoassay within 3 months of recruitment.
- 5. History of at least ≥ 2 recurrent CDI within 6 months where recurrence is defined as return of diarrhea consistent with CDI within 8 weeks following CDI symptom resolution for at least 24 hours after a minimum of 10-day course of standard antibiotic therapy and positive stool test for *C. difficile* toxin or toxin gene and/or ongoing symptoms consistent with CDI despite at least 5 days of treatment using oral vancomycin.
- 6. Has more than three unformed bowel movements or ≥ 200 mL of stool for individuals with a stool collection device such as rectal tube or colostomy during a 24-hour period at the time of initiation of fidaxomicin. Participants will be enrolled when they meet inclusion criteria 1 − 5; will be initiated on fidaxomicin when they have CDI symptoms and stool will be tested for *C. difficile* toxin/gene. Only those with positive stool for *C. difficile* toxin/gene with current episode of CDI will continue with the study
- 7. Females of child bearing potential must be willing to use acceptable birth control as per the Health Canada Guidance Document: Considerations for Inclusion of Women in Clinical Trials and Analysis of Sex Differences.

## 4.2.2 EXCLUSION CRITERIA

- 1. Planned or actively taking an investigational product for another study.
- 2. Prior fidaxomicin use.
- 3. Hypersensitivity to fidaxomicin or to any ingredient in the formulation or component of the container.
- 4. Evidence of toxic megacolon or gastrointestinal perforation or life expectancy of less than 72 hours.
- 5. Active gastroenteritis due to Salmonella, Shigella, E. coli 0157H7, Yersinia or Campylobacter.
- 6. Anticipated requirement for systemic antibiotic therapy for more than 7 days during the study period.
- 7. Actively taking Saccharomyces boulardii or other probiotics other than yogurt.
- 8. Any condition that, in the opinion of the investigator, that the treatment may pose a health risk to the subject.
- 9. Pregnant or lactating.

#### 4.3 SAMPLE SIZE

#### 4.3.1 NUMBER OF SUBJECTS TO BE ENROLLED

A sample size of 50 is planned.

Date: 01OCT2020 

## 4.4 SCREENING, RANDOMIZATION, BLINDING

## 4.4.1 SCREENING PROCEDURE

Potential participants will be screened for eligibility based on the inclusion and exclusion criteria when the PI receives consultation request for recurrent CDI.Patients will be recruited to participate in the trial when they meet the inclusion criteria (1 to 5) and do not have any exclusion ones. The eligible participants with active diarrhea with clinical criteria for CDI will be initiated on fidaxomicin. For those without diarrhea at baseline will be instructed to phone the research office when they experience recurrent symptoms consistent with their previous episodes of CDI. They will be assessed within 48 hours of symptom onset and will be started on fidaxomicin if they continue to meet the inclusion criteria and do not have any exclusion ones. The stool sample collected during the onset of this particular CDI episode will be tested for *C. difficile* toxin. If positive then they will complete the 30-day course of fidaxomicin. If the stool tested negative for *C. difficile* toxin then they will be excluded from further participation of this study and standard of care for this particular episode of diarrhea will be provided based on the most likely etiology.

Females of child bearing potential must be willing to use contraception methods of birth control to participate in the study. Highly effective methods may include: hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation. Highly effective methods of contraception might not always be achievable in the clinical trial setting and, therefore, the most effective alternative can be achieved using methods in combination. Effective methods may include: barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge).

Use of therapeutic products where the risk of fetal abnormality is not known or is unclear (e.g. lack of adequate reproduction toxicity data), animal studies have failed to reveal evidence of fetal harm and use of fidaxomicin, however there are no controlled data in human pregnancy: therefore at least one highly effective method of contraception or two forms of effective contraception methods need to be used.

The half-life of fidaxomicin is 11.7 +/- 4.8 hours therefore will specify to continue with contraception for 48 hours after the last dose of fidaxomicin.

# 4.5 REGULATORY AND ETHICS

#### 4.5.1 INFORMED CONSENT

Informed consent will be obtained from each participant.

## 4.5.2 INSTITUTIONAL REVIEW BOARD/ETHICS COMMITTEE

The study protocol and informed consent form and amendments will be submitted to the Vancouver Island Health Authority Clinical Research Ethics Board.

# 4.5.3 INVESTIGATIONAL NEW DRUG (IND) FILING

No Objection Letter will be obtained from Health Canada.

Date: 01OCT2020 

# 5 STUDY PROCEDURES

# **5.1 TREATMENT**

Participants will take fidaxomicin 200 mg by mouth (PO) twice daily for 10 days, followed by 200 mg PO once daily for 20 days.

# 5.2 STUDY PROCEDURES SCHEDULE

| | Baseline/Day 1 | Unscheduled visit | Day 10 (-3 to +1d) | Week 3 to 12 |
|---|---|---|---|---|
| Procedure | Eligibility screen Obtain consent Medical and CDI history Physical examination Laboratory testing if active diarrhea | Active diarrhea<br>consistent with CDI,<br>collect stool sample<br>and bring to clinic | | Weekly phone |
| Laboratory<br>Testing | CBC, chemistry, creatinine, albumin, sodium, potassium, chloride, alanine transaminase, alkaline phosphatase, bilirubin Stool testing for CD toxin Pregnancy test for females of child bearing potential | CBC, chemistry, creatinine, albumin, sodium, potassium, chloride, alanine transaminase, alkaline phosphatase, bilirubin Stool testing for CD toxin, only if active diarrhea | CBC, chemistry, creatinine, albumin, sodium, potassium, chloride, alanine transaminase, alkaline phosphatase, bilirubin | call |

Date: 01OCT2020 

#### 5.3 STUDY TREATMENT SCHEDULE

| | Day 1 to 10 | Day 11 to 30 |
|---|---|---|
| Treatment | Fidaxomicin 200mg by<br>mouth twice daily for 10<br>days | Fidaxomicin 200mg by mouth once daily for 20 days |

# 6 SERIOUS ADVERSE DRUG REACTIONS

#### 6.1.1 **DEFINITONS**

Each serious adverse drug reaction (SADR) which is subject to expedited reporting to Health Canada should be reported individually in accordance with the data element(s) specified in the Health Canada/ICH Guidance Document E2A: "Clinical Safety Data Management: Definitions and Standards for Expedited Reporting". Expedited reports are required for events that meet all of these three criteria: serious, unexpected and a suspected causal relationship.

**Serious**: Any untoward medical occurrence that at any dose:

- Results in death
- Life-threatening
- Requires inpatient hospitalisation or prolongation of existing hospitalisation
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect.

# 6.1.2 RELATIONSHIP TO STUDY MEDICATION

Event reaction causality scoring system will be used to determine the probability of relationship to study medication

## 6.1.3 EXPECTEDNESS OF ADR

An "unexpected" adverse reaction is one in which the nature or severity is not consistent with information in the relevant source document(s), such as the IB or Product Monograph.

## 6.1.4 RECORDING AND REPORTING SADR

SADRs which are unexpected, serious AND suspected causal relationship to the study medication will be reported to the research ethics board within 24 hours of the PI being aware of the event. This information will also be reported to Health Canada:

Health Canada Office of Clinical Trials

Protocol No: CDI.FIDAXOMICIN.1 Version No. 5 Date: 01OCT2020  Therapeutic Products Directorate 5th Floor, Holland Cross, Tower B A/L 3015A 1600 Scott Street Ottawa, Ontario Canada K1A 0K9

Fax: 613-941-2121

# 7 DATA COLLECTION AND ANALYSIS

## 7.1 DATA COLLECTION

Data will be collected at baseline, at initiation of fidaxomicin, on day 10, day 30 and 8 weeks post treatment (week 12 of study) using source documents

## 7.2 DATA VALIDATION

All data collected during the study will be validated by a second research staff using the investigator's clinical notes, electronic medical records, and laboratory results comparing to the source documents

#### 7.3 DATA / STATISTICAL ANALYSIS

The clinical cure rate will be determined using standard binary outcome protocols. Also, logistic regression and survival analysis methods will be performed. The primary endpoints of clinical response, sustained clinical response, time to resolution of diarrhea (TTROD), recurrence of CDI, and treatment failure will be analyzed by logistical regression.

# **8 PUBLICATION**

The abstract will be submitted for presentation at Infectious Diseases Society of America or Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC). The manuscript will be submitted to a medical journal.

# 9 REFERENCES

- 1. Kelly CP, LaMont JT *Clostridium difficile*-more difficult than ever. *N Engl J Med* 2008;359:1932-40.
- 2. Loo VG, Poirier L, Miller MA, et al. A predominantly clonal multi-institutional outbreak of *Clostridium difficile* -associated diarrhea with high morbidity and mortality. *N Engl J Med* 2005;353:2442-9.
- 3. Lavallée C, Laufer B, Pépin J, Mitchell A, Dubé S, Labbé AC. Fatal *Clostridium difficile* enteritis caused by the BI/NAP1/027 strain: a case series of ileal *C. difficile* infections. *Clin Microbiol Infect* 2009:15:1093-9.
- 4. O'Connor JR, Johnson S, Gerding DN. *Clostridium difficile* infection caused by the epidemic BI/NAP1/027 strain. *Gastroenterology* 2009;136:1913-24.
- 5. Quesada-Gómez C, Rodríguez C, Gamboa-Coronado Mdel M, Rodríguez-Cavallini E, Du T, Mulvey MR, Villalobos-Zúñiga M, Boza-Cordero R. Emergence of *Clostridium difficile* NAP1 in Latin America. *J Clin Microbiol* 2010;48:669-70.
- 6. Pillai DR, Longtin J, Low DE. Surveillance data on outbreaks of *Clostridium difficile* infection in Ontario, Canada, in 2008-2009. *Clin Infect Dis* 2010;50:1685-1686.

Date: 01OCT2020 

- 7. Vonberg RP, Reichardt C, Behnke M. et. al. Cost of nosocomial *Clostridium difficile*-associated diarrhea. *J Hosp Infect* 2008;70:15-20.
- 8. Dubberke ER, Olsen MA. Burden of *Clostridium difficile* on the healthcare system. *Clin Infect Dis* 2012;55(suppl 2): S88-92.
- 9. O'Horo JC, Jindai K, Kunzer B, Safdar N. Treatment of recurrent *Clostridium difficile* infection: a systematic review. *Infection*. 2014;42(1):43-59. doi:10.1007/s15010-013-0496-x.
- 10. Petrella L a., Sambol SP, Cheknis A, et al. Decreased cure and increased recurrence rates for clostridium difficile infection caused by the Epidemic *C. difficile* BI strain. *Clin Infect Dis*. 2012;55(3):351-357. doi:10.1093/cid/cis430
- 11. Pépin J, Saheb N, Coulombe M-A, et al. Emergence of fluoroquinolones as the predominant risk factor for Clostridium difficile-associated diarrhea: a cohort study during an epidemic in Quebec. *Clin Infect Dis.* 2005;41(9):1254-1260.
- 12. McFarland L V., Elmer GW, Surawicz CM. Breaking the cycle: Treatment strategies for 163 cases of recurrent Clostridium difficile disease. *Am J Gastroenterol*. 2002;97(7):1769-1775.
- 13. van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. *N Engl J Med.* 2013 Jan 31;368(5):407-15.
- 14. Guo B, Harstall C, Louie T, Veldhuyzen van Zanten S, Dieleman L. Systematic review: faecal transplantation for the treatment of *Clostridium difficle*-associated disease. *Aliment Pharmacol Ther* 2012;35:865-875.
- 15. Gough E, Shaikh H, Manges AR. Systematic Review of Intestinal Microbiota Transplantation (Fecal Bacteriotherapy) for Recurrent *Clostridium difficile* Infection. *Clin Infect Dis* 2011;53(10):994-1002.
- 16. Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. *Am J Gastroenterol*. 2013;108(4):500-8. doi:10.1038/ajg.2013.59.
- 17. Louie T, Miller M, Mullane K, Weiss K, Lentnek A. et.al. Fidaxomicin versus Vancomycin for *Clostridium difficile* infection. *N Engl J Med* 2011;364:422-31.
- 18. Louie T, Emery J, Krulicki W, Byrne B, Mah M. OPT-80 Eliminates *Clostridium difficile* and Is Sparing of *Bacteroides* Species during Treatment of *C. difficile* Infection. Antimicrob. Agents Chemother 2009;53: 261-263.
- 19. Health Canada Guidance Document For Clinical Trial Sponsors: Clinical Trial Applications dated May 29, 2013. Available at: http://www.hc-sc.gc.ca/dhp-mps/prodpharma/applic-demande/guide-ld/clini/ctdcta ctddec-eng.php. Accessed 2015-Feb-18.
- 20. Health Canada Guidance Document: Considerations for Inclusion of Women in Clinical Trials and Analysis of Sex Differences. Appendix A: Considerations in using contraceptives in clinical trials. Dated May 29, 2013. Available at: http://www.hc-sc.gc.ca/dhp-mps/prodpharma/applic-demande/guide-ld/clini/womct\_femec-eng.php#aa. Accessed 2015-Feb-18.

Date: 01OCT2020 

Protocol No: CDI.FIDAXOMICIN.1 Date: 01OCT2020

# **Appendix A: Telephone Script**

| PHONE CONTACT SCHEDULE AND SCRIPT Weekly contact by phone –Week 3 to 8 | |
|---|---|
| Participant phone follow-up script: | |
| Participant ID: | |
| Date:// | Time::: |
| Mr./Mrs./Mstreatment of <i>Clostridioides difficile</i> | from Vancouver Island Health Authority. I would like to speak to in regards to his/her participation in the research study for the infection. Mr./Mrs./Ms, May I ask you a couple articipation in this study? All of the information that you share with |
| Daily contact in person or by pho | ne: |
| <ol> <li>How has your overall healt</li> <li>Have you experienced any</li> </ol> | been since we last spoke? Informed bowel movement since we last spoke? Yes/No |

If yes, have you had three or more unformed bowel movements in any 24 hour period during the follow-up? If yes, you will need to return for assessment, bloodwork and stool collection.

Thank you for your time and your participation in this important research project.

Date: 01OCT2020 